CLINICAL TRIAL: NCT02202707
Title: Vasomotor Symptoms and Cardiovascular Control
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: No funding obtained to conduct study
Sponsor: Beth Israel Deaconess Medical Center (Other)
Collaborators: Brigham and Women's Hospital (Other); Spaulding Rehabilitation Hospital (Other)
Responsible Party: Principal Investigator, Suzanne Bertisch, BIDMC Site Investigator, Beth Israel Deaconess Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2013P002024
Record Dates: First submitted 2014-07-22; First posted 2014-07-29 (Estimated); Last update posted 2015-08-19 (Estimated); Status verified 2015-08

CONDITIONS: Vasomotor Symptoms; Cardiovascular Health
MeSH Terms: interventions — Gabapentin

ARMS (1):
- Gabapentin (Other): Open label single arm study. All participants will receive Gabapentin.
  Interventions: Drug: Gabapentin

INTERVENTIONS:
Drug: Gabapentin — Study medication, gabapentin, will be distributed to all study participants and participants will be instructed as to how to take and titrate the medication dose. Participants will take gabapentin daily for up to six weeks.
  Other Names: Neurontin

SUMMARY:
The purpose of this study is to preliminarily determine whether the frequency and/or severity of vasomotor symptoms (VMS) at baseline, and then after symptom reduction with gabapentin, relates to various cardiovascular control measures.

DETAILED DESCRIPTION:
Visit 1: Screening & Acclimation Visit

The informed consent process for the study will be completed and a signed informed consent form will be obtained at Spaulding Hospital Cambridge. Subjects will be screened to ensure they meet preliminary eligibility criteria. All subjects will undergo a clinical interview to determine the presence of any medical disorders. The following study assessments will be completed:

* 12-lead EKG
* Resting blood pressure and heart rate
* Height and Weight

Visit 2: VMS Determination and At-Home Assessments Subjects will be interviewed about their mental health history, and will complete questionnaires about their VMS, related quality-of-life symptoms (sleep, mood) and quality-of-life. Blood will be drawn to confirm eligibility and to assess for diabetes and chronic kidney disease (see exclusion criteria). Subjects will be given a 7-day VMS Diary and a 7-day Sleep Diary at the end of this visit, to be completed at home during the following week. Participants will also be given an actigraphic watch to take home to wear for 7 days in order to capture sleep/wake patterns and activity levels for exploratory analyses. During the 7 days of at-home VMS and sleep monitoring, subjects will also wear a portable VMS monitor for 24 hours to measure objective VMS frequency.

Visit 3: Final Eligibility Determination & Lab VMS Monitoring Subjects will return the objective VMS monitor and the VMS and sleep diaries, and the results of their blood tests taken during the Visit 2 will be reviewed to ensure eligibility. Eligible subjects will participate in a 6-hour laboratory objective VMS monitoring session by wearing an objective VMS monitor while simultaneously subjectively monitoring VMS experienced with a written diary and an event marker. Objective VMS measures obtained during this visit will be the primary baseline measure of VMS for investigation. Those who have at least 2 objective VMS measured during the 6-hour monitoring period will be deemed eligible and referred for baseline studies and to start medication. Participants will be given additional VMS and sleep diaries to complete on a daily basis throughout the rest of the study period.

Visit 4: Laboratory Testing Visit & Medication Distribution All studies will be performed between ~8-10 am and will occur at the same time for the second laboratory testing visit. All subjects will be instructed to abstain from vigorous exercise for 2 days prior to each study to avoid autonomic and neuroendocrine effects of exercise. In addition, subjects will refrain from caffeine and alcohol for the previous 24 hrs, and be studied after a 12 hr fast.

A. Study Visit: Parameters to be Measured

1. Electrocardiogram.
2. Arterial Pressure.
3. Respiration.
4. Sympathetic Microneurography.
5. Beat-by-Beat Leg Blood Flow. B. Drugs to Study Human Physiology

1) Intravenous bolus injection of 100 ug nitroprusside bolus (a vasodilator which drops pressure) 2) Intravenous bolus injection 150 ug phenylephrine bolus (a vasoconstrictor which raises pressure).

These two drugs are used to drop and raise pressure through a range of arterial pressures within a very short time, approximately 2 minutes.

These medications raise and lower blood pressure by the same amount typically experienced during the day when performing activities such as climbing stairs or moving from sitting to standing.

C. Data to be collected/Timing of collection The study visit will take about 4 hours. Throughout the protocol, subjects will lie supine and will be instrumented for measurement of the ECG, beat-by-beat arterial pressure, brachial arterial pressure, respiratory excursions, and popliteal blood flow velocity. After instrumentation and calibration, instrumentation for measurement of peroneal nerve muscle sympathetic activity will commence, with the internal search lasting a maximum of 60 minutes.

After either successful or unsuccessful procurement of the nerve recording, the testing protocol will start:

Testing Protocol

1. Baseline recordings/measurement (~10 minutes): Subjects will rest quietly for 10 minutes.
2. Modified Oxford Baroreflex tests (5 minutes/trial, 2 trials, ~30 minutes total): An intravenous bolus injection of 100 ug nitroprusside bolus, followed in 1 minute by a 150 ug phenylephrine bolus. After the first trial, a second modified Oxford baroreflex test will be performed. At least 10-15 minutes will be allowed between the baroreflex trials to insure that heart rate, blood pressure and nerve activity return to resting levels. Subjects will be continually assessed for adverse events and symptoms related to hypotension.
3. Sustained isometric handgrip exercise (~10 minutes): Subjects will be asked to perform an isometric handgrip exercise at 30% of maximum effort sustained to fatigue.
4. Valsalva's maneuver (~5 minutes): Subjects will be asked to blow into a tube via a mouthpiece and generate a pressure of ~40 mmHg sustained for 12 seconds. Data will be collected for one minute prior to the maneuver, one minute after, with two minutes of recovery between trials. This will be repeated to obtain three successful trials.
5. Paced breathing (~15 minutes total): Subjects will be asked to maintain a constant breathing frequency of 15 breaths/min (0.25 Hz) following an audio signal (i.e., "in, two, out, two") for 5 minutes after a short period of acclimation.

Distribution of Study Medication: After all baseline measures are complete, study medication (gabapentin) will be distributed to all study participants and participants will be instructed as to how to take and titrate the medication dose.

Visit 5a: Medication Dosage & Adverse Event Monitoring (Telephone) Study staff will check in with study participants over the telephone after they have been on gabapentin for approximately one week to monitor any side effects or adverse events of the medication. If subjects are experiencing intolerable side effects, they will be taken off of the medication while completing the remaining study procedures. In order to track potential after effects of microneurography, subjects who had the electrode placed beneath the surface of their skin will be given the Microneurography Questionnaire (MSNA). Over the last 18 years of performing the technique, roughly 5% of participants have after effects, and of these the most often reported effect (>90%) is slight bruising at the site of insertion.

Visit 5b: Medication Dosage & Adverse Event Monitoring (Telephone) Study staff will check in with study participants over the telephone after they have been on gabapentin for approximately three weeks to monitor any side effects or adverse events of the medication. If subjects are experiencing intolerable side effects, they will be taken off of the medication while completing the remaining study procedures.

Visit 6: Objective VMS Monitoring All subjects will repeat the 6-hour laboratory objective VMS monitoring session on gabapentin for post-treatment measures of VMS, as described above for Visit 3. Participants will also complete the same set of pre-treatment questionnaires about their VMS, related quality-of-life symptoms (sleep, mood) and quality-of-life. All subjects will be given the ambulatory VMS monitor to wear for 24 hours at home, to capture the frequency of VMS in the ambulatory setting as well as the actigraphic watch to wear for a one-week period. Participants will be reminded to continue to complete their VMS and sleep diaries.

Visit 7: Laboratory Testing Visit & Medication Collection Procedures performed during Visit 4 will be repeated at Visit 7, to collect data on cardiovascular measures after participants have been on gabapentin for at least 4 weeks at the full dose. All VMS and sleep diaries, as well as unused study medication, actigraphic watch, and the objective VMS monitor, will be returned and collected at this visit.

ELIGIBILITY:
Inclusion Criteria:

1. Women aged 45 to 58 years,
2. Early postmenopausal, defined as a minimum of one year and up to 6 years from final menstrual period (FMP)
3. Vasomotor symptoms for at least 6 months

   * At least 4/day or 28/week by retrospective report and confirmed on prospective monitoring over 2-week period.
   * At least 2 VMS measured objectively on the VMS monitor during the 6-hour VMS laboratory monitoring session.
4. Normal to overweight (18.5≤BMI≤35 kg/m2)
5. Sedentary to normally physically active (performing regular aerobic exercise <60 min/week)

Exclusion Criteria:

1. Hypertension (resting pressures ≥140/90 mmHg)
2. Diabetes (verified by plasma hemoglobin A1C level ≥6.5)
3. Cardiovascular disease, including any stenotic valvular heart disease
4. Neurological disease
5. Current depression (per screening procedures)
6. Current or history of suicidal ideation or attempts (within 3 years prior to enrollment)
7. Lifetime history of bipolar disorder
8. Active cancer (non-melanoma skin cancer allowed)
9. Abnormal resting ECG
10. Recent weight change (>10 lb weight change in last 6 months)
11. Regular tobacco use/current smoking
12. Current use of anti-hypertensives or other medications that could influence any of the dependent variables
13. Current or previous use (past 2 months) of anti-anxiety, anti-depressant or antipsychotic medications
14. Current use of vasodilators
15. Current use of stimulants or stimulant-like medications
16. Current use of systemic hormone therapies/medications
17. Current use of non-hormonal treatments for VMS
18. Current use of gabapentin or medications contraindicated to be used in combination with gabapentin
19. Past intolerance or hypersensitivity to gabapentin
20. History of syncope or vasovagal/carotid sensitivity
21. History of sickle cell anemia
22. Abnormal kidney function: CrCl or GFR <60 ml/min (Cockcroft and Gault equation)
23. Ventricular tachycardia
24. Hyperthyroidism
25. Hypersensitivity to phenylephrine
26. Compensatory hypertension, where the primary hemodynamic lesion is aortic coarctation or arteriovenous shunting
27. Congenital (Leber's) optic atrophy or tobacco amblyopia
28. Hypersensitivity to nitroprusside

Ages: 45 Years to 58 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2014-05; Primary Completion 2016-06 (Estimated); Study Completion 2016-06 (Estimated)

PRIMARY OUTCOMES:
Alterations in cardiovagal tone with treatment of vasomotor symptoms in women | 5 weeks
  Cardiovagal tone will be assessed using heart rate and blood pressure at rest and in response to pharmacological and physical tasks
Alterations in sympathetic efferent outflow with treatment of vasomotor symptoms | 5 weeks
  muscle sympathetic nerve activity at rest and in response to pharmacological and physical tasks

CONTACTS AND LOCATIONS:
Overall Officials: J. Andrew Taylor, PhD, Principal Investigator — Spaulding Hospital Cambridge
Locations (2):
- United States (2):
  - Brigham and Women's Hospital, Boston, Massachusetts
  - Spaulding Hospital Cambridge, Cambridge, Massachusetts